CLINICAL TRIAL: NCT07249385
Title: Nudging Provider Adoption of Clinical Decision Support: Implementation of an EHR-Agnostic Pulmonary Embolism Risk Prediction Tool
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-01528; 5R01HL169364-02 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Compact Disks; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Each emergency department (ED) will function as a control group (usual care) prior to implementation of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Department (ED) Providers (Experimental): Each ED will serve as its own control. Baseline data will be collected for 12 months prior to the implementation of the CDS system with nudges. The CDS tool with nudges will then be implemented for 33 months.
  Interventions: Behavioral: Clinical Decision Support (CDS) tool with Nudges

INTERVENTIONS:
Behavioral: Clinical Decision Support (CDS) tool with Nudges — The CDS tool with nudges provide information to providers to practice medicine in accordance with CT (computed tomography) ordering guidelines. The tool will only deploy when the provider is going against clinical guidelines and therefore provides a chance for the provider to reconsider their actions.

SUMMARY:
The purpose of this study is to examine the impact of the nudge implementation strategy (CDS tool + Nudge) on adoption of guideline-concordant CT ordering for pulmonary embolism (PE) in 10 EDs. The study will be a 33-month, rigorous, pragmatic, cluster-randomized, stepped wedge trial across 3 health systems and 10 EDs after collecting pre-implementation baseline data. The aim is to to demonstrate technological feasibility as well as examine efficacy of the nudges on adoption. The secondary objective is to decrease CT-ordering when it is not indicated.

DETAILED DESCRIPTION:
Part 1 of the study included the collection of data. During the pre-implementation period each sites electronic health record (EHR) and baseline data was collected for 12 months. In Part 2, the study will examine the impact of the nudge implementation strategy (CDS tool + Nudge) on adoption of guideline-concordant CT ordering for PE in 10 EDs. Adoption outcomes data will be collected through EHR reporting systems.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of older
2. A provider (MD, NP, PA) ordering CTs for evaluation of PE in adult patients present at study site Emergency Department (i.e., Northwell Health - Feinstein Institute for Medical Research, Baylor College of Medicine and NYU Langone Health).

Exclusion Criteria:

1. A provider not present at the specified study sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of CT scan orders that are guideline-concordant | Baseline (Month 12)
  Guideline-concordant is defined as CT scan orders with Wells' Score >4 ["PE Likely"] and/or d-dimer above upper limit of normal.
Percentage of CT scan orders that are guideline-concordant | End of intervention (Month 45)
  Guideline-concordant is defined as CT scan orders with Wells' Score >4 ["PE Likely"] and/or d-dimer above upper limit of normal.

CONTACTS AND LOCATIONS:
Overall Officials: Safiya Richardson, MD MPH, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Northwell Health - Feinstein Institute for Medical Research, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Safiya.richardson@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Safiya.richardson@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.